CLINICAL TRIAL: NCT06104189
Title: Ultrafast MRI Radiomics to Classify Histological Factors and Subtypes of Breast Cancer
Brief Title: Prospective Ultrafast MRI Radiomics for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Bo Kyoung Seo, Professor, Korea University Ansan Hospital
Other Study IDs: UFMRIRADIOMICS
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — MRI based classification of breast cancer histological factors and subtypes

SUMMARY:
The goal of this prospective study is to investigate the performance of ultrafast MRI radiomics in classifying histological factors and subtypes of breast cancer compared with standard MRI among radiologists with varying experience. The written informed consent was obtained from all participant. We extracted 1618 radiomic features from ultrafast and standard contrast-enhanced MRI before treatment. Classification of hormonal receptors, human epidermal growth factor receptor 2, and Ki67 status and subtypes was evaluated using the area under the receiver-operating characteristic curve (AUC) with the DeLong test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with invasive breast cancer

Exclusion Criteria:

* Diagnosed with other cancer

Ages: 27 Years to 86 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population should fulfill the following criteria as follows:(a) histologically confirmed invasive breast cancer, (b) participant consent, and (c) MRI performed before treatment.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The signal intensity of MRI according to histological factors and subtypes of breast cancer | Baseline, pre-surgery
  Quantitative image values obtained from ultrafast MRI show similar performance in classifying histological factors and subtypes compared with standard MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Kyoung Seo, MD, PhD, Principal Investigator — Korea University Ansan Hospital
Locations (1):
- Bo Kyoung Seo, Ansan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jeong J, Ham S, Seo BK, Lee JT, Wang S, Bae MS, Cho KR, Woo OH, Song SE, Choi H. Superior performance in classification of breast cancer molecular subtype and histological factors by radiomics based on ultrafast MRI over standard MRI: evidence from a prospective study. Radiol Med. 2025 Mar;130(3):368-380. doi: 10.1007/s11547-025-01956-6. Epub 2025 Jan 25. PMID 39862364